CLINICAL TRIAL: NCT02447692
Title: Proportional Assist Ventilation for Minimizing the Duration of Mechanical Ventilation: The PROMIZING Study
Acronym: PROMIZING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Medtronic (Industry); Canadian Critical Care Trials Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPR-327433, ISR-2014-10481
Record Dates: First submitted 2015-05-08; First posted 2015-05-19 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2024-08

CONDITIONS: Critically Ill; Acute Respiratory Failure
Keywords: Proportional Assist Ventilation; Pressure Support Ventilation; Weaning
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSV ventilation strategy (Active Comparator): The control is the standard of care PSV ventilation strategy, designed to adjust the level of support according to usual clinical parameters.
  Interventions: Other: PSV ventilation strategy
- PAV+ ventilation strategy (Active Comparator): The intervention is a PAV+ ventilation strategy, designed to adjust the level of support (gain) to target a predefined range of respiratory muscle pressure.
  Interventions: Other: PAV+ ventilation strategy

INTERVENTIONS:
Other: PSV ventilation strategy — An algorithm for adjusting the level of pressure support according to usual clinical parameters; patients not tolerating PSV will be switched to Assist/Control mode according to predefined criteria
  Arms: PSV ventilation strategy
Other: PAV+ ventilation strategy — An algorithm for adjusting the level of support (gain) to maintain a predefined range of respiratory muscle pressure; patients not tolerating PAV+ (Puritan Bennett™ 840 or 980 ventilator) will be switched to Assist/Control mode according to predefined criteria
  Arms: PAV+ ventilation strategy

SUMMARY:
For adult patients with acute respiratory failure requiring invasive mechanical ventilation, does a ventilation strategy using proportional assist ventilation with load-adjustable gain factors (PAV+) result in a shorter duration of time spent on mechanical ventilation than a ventilation strategy using pressure support ventilation (PSV)?

DETAILED DESCRIPTION:
Patients with acute respiratory failure require mechanical ventilation to help them breathe until they recover from their acute illness. Although mechanical ventilation is necessary to sustain life in such situations, it can induce weakness of the respiratory muscles which may lead to prolonged dependence on the ventilator. Prolonged dependence on mechanical ventilation is associated with increased mortality, morbidity and costs to the healthcare system. Thus, a main goal of assisted mechanical ventilation is to reduce the patient's respiratory distress while maintaining some respiratory muscle activity. To attain this goal, the amount of ventilator assistance should theoretically be adjusted to target normal or reasonable levels of respiratory effort.

Modes of Mechanical Ventilation:

Proportional assist ventilation with load-adjustable gain factors (PAV+) is a mode of mechanical ventilation which delivers assistance to breathe in proportion to the patient's effort. The proportional assistance, called the gain, can be adjusted by the clinician to maintain the patient's respiratory effort or workload within a reasonable range. This is the only mode of ventilation which allows for measurement and targeting of a specific range of respiratory muscle activity by the patient.

Pressure support ventilation (PSV) is a mode of ventilation which is considered the current standard of care for assisting breathing of patients during the recovery phase of acute respiratory failure. Several studies have shown short term advantages of PAV over PSV, including improved patient-ventilator synchronization, improved adaptability to changes in patient effort, and improved sleep quality.

Goal of this Randomized Controlled Trial:

To demonstrate that for patients with acute respiratory failure, ventilation with PAV+, being more physiological, will result in a shorter duration of time spent on mechanical ventilation than ventilation with PSV.

ELIGIBILITY:
A staged enrolment process will be used to identify patients eligible to be enrolled and randomized in the study. At each stage of the enrolment process, a patient must meet inclusion criteria and not meet exclusion criteria in order to pass. To progress to the next stage, patients must continue to pass criteria from the prior stages. After enrolment, there are also specific tests to perform (with pass/fail criteria) to determine eligibility to be randomized.

A. SCREENING INCLUSION CRITERIA:

* A1. Age 18 years or older
* A2. Intubated and receiving any mode of invasive mechanical ventilation ≥ 24 hours

A. SCREENING EXCLUSION CRITERIA:

* A3. Anticipating withdrawal of life support and/or shift to palliation as the goal of care
* A4. Severe central neurologic disorder (eg. Hemorrhage, stroke, tumour) causing elevated intracranial pressure, or impaired control of breathing, or requiring specific ventilator adjustments (i.e. To attain specific CO2 target) or requiring neurosurgical intervention
* A5. Known or suspected severe or progressive neuromuscular disorder likely to result in prolonged or chronic ventilator dependence (eg. Guillain-Barré syndrome, Myasthenia Gravis, ALS, MS, high spinal cord injury, kyphoscoliosis or other restrictive disorder) (Note that obesity hypoventilation syndrome that may be managed with nocturnal non-invasive ventilation is NOT an exclusion under A5)
* A6. Severe COPD: Baseline daytime hypercapnia (pCO2> 50 mmHg) OR GOLD 4 airflow limitation (FEV1<30% predicted) OR MRC class 4 symptoms ("I am too breathless to leave the house" OR "I am breathless when dressing")
* A7. Broncho-pleural fistula
* A8. Tracheostomy present at ICU admission for the purpose of chronic or prolonged mechanical ventilation (>21 days). (Note that a patient who was endotracheally intubated for acute respiratory failure and received a tracheostomy during their ICU admission, prior to enrolment, is not excluded under A8).
* A9. Current enrolment in a confounding study, as assessed by the steering committee
* A10. Previous randomization in the PROMIZING Study
* A11. Severe, end-stage, irreversible respiratory or cardiac disease (e.g. interstitial lung disease, pulmonary fibrosis, cardiomyopathy, valvulopathy) likely to result in prolonged or chronic ventilator dependence /unlikely to wean from mechanical ventilation [Note: patients who are candidates for intervention to treat the underlying respiratory/cardiac disease (e.g. lung transplant, heart transplant, cardiac surgery) may be re-evaluated once intervention is complete and they no longer meet criteria A11.]

B. ENROLMENT INCLUSION CRITERIA:

* B1. Ability or potential ability to trigger ventilator breaths (i.e. not receiving neuromuscular blockade).
* B2. On Assist/Control volume-cycled ventilation: Technically satisfactory plateau pressure ≤ 30 cm H2O (see Operations Manual) OR On Assist/Control pressure-controlled ventilation or similar mode: Pressure control plus PEEP ≤ 30 cm H2O OR On Pressure Support ventilation: Pressure support plus PEEP ≤ 30 cm H2O OR On Proportional Assist ventilation: PAV gain <85%
* B3. PaO2 ≥ 60 mmHg or SpO2 ≥ 90% on FiO2 ≤ 0.60 and PEEP ≤ 15 cm H2O
* B4. Metabolic disorders corrected: pH ≥7.32
* B5. Stable hemodynamic status: stable or decreasing doses of vasopressors for ≥6 hours
* B6. Anticipate ongoing need for ventilation >24 hours

B. ENROLMENT EXCLUSION CRITERIA:

* B7. Extubated
* B8. Died
* B9. Patient has met enrolment inclusion criteria B1-B5 AND has tolerated pressure support of 0-20 cm H2O or proportional assist ventilation of 0-85% for ≥24 consecutive hours (including time on CPAP, t-piece, or tracheostomy mask). (Note (1): that it is acceptable to include a patient who has been tried on pressure support or proportional assist ventilation but has required pressures >20 cmH2O or assistance >85% or has required return to A/C ventilation within the 24 hour time window; Note (2): B9 does not apply to patients on ECMO.)
* B10. Patient transferred to a non-participating centre

B. ENROLMENT DEFERRAL CRITERIA:

* B11. Plan to extubate/discontinue mechanical ventilation within <24 hours (Reassess within 24 hours)
* B12. Patient currently on ECMO (Reassess patient once off ECMO)
* C9: Plan for surgery or complex procedure that will require full ventilation to be done prior to attempting extubation (e.g. Procedure requiring neuromuscular blockade and/or heavy sedation, such that patient would be apneic, or not be able to trigger ventilator) (Reassess after surgery/procedure complete)

C. PRESSURE SUPPORT TRIAL INCLUSION CRITEIRA:

* C2. Upon review of Screening and Enrolment criteria (A and B), the patient still passes.
* C3. Treating physician has provided verbal consent to proceed with standardized tests and randomization if eligibility criteria are met.

C. PRESSURE SUPPORT TRIAL DEFERRAL CRITERIA:

* C6. High dose vasopressor requirements (i.e. epinephrine or norepinephrine >0.5 ug/kg/min or equivalent) OR patient requiring an increase in dose of vasopressor within 6 hrs
* C7. Active cardiac ischemia (dynamic ST changes on monitor or ECG within 6 hours)
* C8. Unstable arrhythmias (HR>140 or <50) with clinical signs of low cardiac output or or SBP<80 mmHg
* C10. Receiving a "strict lung protective" ventilation strategy for ARDS (eg. Order on chart to keep Vt ≤6 mL/kg PBW)

C. PRESSURE SUPPORT TRIAL EXCLUSION CRITERIA:

• C12. Treating physician has declined consent

D. WEANING CRITERIA:

* D1. SpO2≥ 90% on FiO2 ≤0.40 and PEEP ≤8 cmH2O
* D2. pH ≥7.32
* D3. Vasopressor requirements no higher than norepinephrine 0.1 ug/kg/min or equivalent.

In the final stage (E), patients will be considered eligible for randomization if the following criteria are met.

E. RANDOMIZATION INCLUSION CRITERIA:

* C1. Patient/SDM has provided consent OR Plan to obtain deferred consent as Patient incapable and no SDM available to provide consent within the randomization window
* E1. Upon review of Criteria A, B, and C, the patient still passes and the patient has passed the PST.
* E2. Does not meet Weaning Criteria OR Fails the ZERO CPAP Trial OR Fails the SBT

E. RANDOMIZATION EXCLUSION CRITERIA:

* B9. Patient has met enrolment inclusion criteria B1-B5 AND has tolerated pressure support of 0-20 cm H2O or proportional assist ventilation of 0-85% ≥24 consecutive hours (including time on CPAP, t-piece, or tracheostomy mask). Note (1): It is acceptable to include a patient who has been tried on pressure support or proportional assist ventilation but has required pressures >20 cmH2O or assistance >85% or has required return to A/C ventilation within the 24 hour time window; Note (2): B9 does not apply to patients while on ECMO
* C4. Patient/SDM has declined consent
* C5. Patient incapable and no SDM available to provide consent (not applicable if plan to obtain deferred consent)
* E3. Passed SBT on t-piece, FiO2 0.40 for 30-120 minutes
* E4. Approval withdrawn (by physician or patient/SDM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Time from randomization to successful liberation from invasive mechanical ventilation. | up to 90 days
  "Successful liberation" is defined as removal of the endotracheal tube AND remaining alive with no need for reintubation/reinstitution of invasive mechanical ventilation for 7 days post extubation, or until successful ICU discharge, or until live hospital discharge, whichever comes first.

SECONDARY OUTCOMES:
Ventilator-free days at 14, 21 and 28 days post randomization | 14, 21 and 28 days post randomization
  "Ventilator-free days" (VFDs) are defined as the number of days alive and free of INVASIVE ventilation post SUCCESSFUL EXTUBATION or post successful termination of invasive mechanical ventilation (MV) from time of randomization to day 21 post randomization. "Successful extubation" is defined as removal of the endotracheal tube AND remaining alive with no need for reintubation/reinstitution of invasive mechanical ventilation for 7 days post extubation, or until successful ICU discharge, or until live hospital discharge, whichever comes first.
Time from randomization to live ICU discharge (up to day 90) | up to 90 days
  Patients will remain in the study and will continue on the assigned ventilation strategy until: successful extubation, successful ICU discharge, live hospital discharge, death, or 90 days post randomization, whichever comes first.
Time from randomization to live hospital discharge (up to day 90) | up to 90 days
  Patients will remain in the study and will continue on the assigned ventilation strategy until: successful extubation, successful ICU discharge, live hospital discharge, death, or 90 days post randomization, whichever comes first.
Mortality | up to 90 days
  Measured as time to death, ICU mortality; hospital mortality; 21, 28, and 90 day mortality
Weaning Progress | up to 90 days
  Measured as time from randomization to: first SBT; first successful SBT; first extubation
Weaning Difficulties | 90 days
  Measured as the number of patients failing first SBT or first extubation attempt and requiring up to 7 days to extubate (difficult weaning group/group 2); failing first SBT or first extubation attempt and requiring more than 7 days to extubate (prolonged weaning group/group 3)
Weaning Complications | 90 days
  Measured as the number of patients: requiring non-invasive ventilation post-extubation; ventilated more than 7 days post randomization, ventilated more than 21 days from time of intubation (prolonged MV group); receiving tracheostomy post-randomization, requiring re-intubation (up to 7d after planned extubation)
Tolerance of modes | 90 days
  Measured as number of patients ever requiring A/C mode post randomization; number of patient-days requiring A/C mode post randomization
Serious Adverse Events | 90 days
  Incidence of reported serious adverse events

OTHER OUTCOMES:
Co-interventions | 28 days
  Co-interventions will be monitored and described including use of sedating medications
Subgroup analyses based on: (a) duration of MV prior to randomization as a continuous variable or as a binary variable of greater than 5 days | At randomization
  Identifies a subgroup of patients at time of randomization who are at risk for prolonged weaning
Subgroup analyses based on (b) failing an SBT prior to randomization vs. failed CPAP 0 trial vs. failed weaning criteria prior to randomization | At randomization
  Identifies a subgroup of patients at time of randomization classified as difficult weaning vs. failed CPAP 0 trial vs. failed weaning criteria prior to randomization
Subgroup analyses based on (c) failed extubation prior to randomization | At randomization
  Identifies a subgroup of patients at time of randomization classified as having "difficult weaning".
Subgroup analyses based on (d) mild vs. moderate vs. severe frailty | At ICU admission
  Differentiates between severely frail and less frail
Subgroup analyses based on COVID-19 positive test | At ICU admission
  Differentiates between COVID-19 positive and COVID-19 negative
Subgroup analyses based on tracheostomy present at randomization | At randomization
  Identifies a subgroup of patients at risk of prolonged weaning

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Bosma, Principal Investigator — London Health Sciences Centre, London, Ontario, Canada; Laurent Brochard, Principal Investigator — St. Michael's Hospital, Toronto, Ontario, Canada
Locations (22):
- El Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno", Buenos Aires, Argentina
- Canada (11):
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Sunnybrook Hospital - Health Sciences Centre, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - UHN- Toronto General Hospital, Toronto, Ontario
  - UHN- Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
- France (5):
  - Centre Hospitalier Universitaire (CHU) de Angers, Angers
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Henri Mondor (Assistance Publique-Hôpitaux de Paris), Créteil
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Centre Hospitalier Universitaire (CHU) de Rouen, Rouen
- University Hospital of Heraklion, Heraklion, Greece
- Italy (2):
  - University Hospital of Ferrara, Ferrara
  - San Giovanni Battista University Hospital, Turin
- King Abdulaziz Medical City, Riyadh, Saudi Arabia
- Hospital de Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected electronically and stored at the Clinical Coordinating Center at the Applied Health Research Centre (AHRC). A de-identified database of all data may be made available for use 3 years after the primary publication upon request and review of the statistical analysis plan by the PROMIZING steering committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after the primary publication

REFERENCES:
- [Derived] Bosma KJ, Burns KEA, Martin CM, Skrobik Y, Mancebo Cortes J, Mulligan S, Lafreniere-Roula M, Thorpe KE, Suarez Montero JC, Moran Chorro I, Rodriguez-Farre N, Butler R, Bentall T, Beduneau G, Enguerrand P, Santos M, Piraino T, Spadaro S, Montanaro F, Basmaji J, Campbell E, Mercat A, Beloncle FM, Carteaux G, Maraffi T, Charbonney E, Lecronier M, Dres M, Arabi YM, Amaral ACK, Marinoff N, Adhikari NKJ, Geagea A, Shin P, Vaporidi K, Kondili E, Shahin J, Campisi J, Rodriguez PO, Setten M, Goligher EC, Ferguson ND, Fanelli V, Ferreyra G, Lellouche F, Sibley S, Brochard L; PROMIZING Study Investigators, the Canadian Critical Care Trials Group, and the REVA Network. Proportional-Assist Ventilation for Minimizing the Duration of Mechanical Ventilation. N Engl J Med. 2025 Sep 18;393(11):1088-1103. doi: 10.1056/NEJMoa2505708. Epub 2025 Jun 13. PMID 40513024
- [Derived] Bosma KJ, Lafreniere-Roula M, Jiang A, Heath A, Ouyang Y, Wade K, Hu P, Burns KEA, Martin CM, Skrobik Y, Mulligan S, Thorpe KE, Brochard L; members of the Canadian Critical Care Trials Group and the REVA Network. Proportional Assist Ventilation for Minimizing the Duration of Mechanical Ventilation (the PROMIZING study): update to the statistical analysis plan for a randomized controlled trial. Trials. 2024 Dec 30;25(1):855. doi: 10.1186/s13063-024-08669-7. PMID 39736673
- [Derived] Bosma KJ, Martin CM, Burns KEA, Mancebo Cortes J, Suarez Montero JC, Skrobik Y, Thorpe KE, Amaral ACK, Arabi Y, Basmaji J, Beduneau G, Beloncle F, Carteaux G, Charbonney E, Demoule A, Dres M, Fanelli V, Geagea A, Goligher E, Lellouche F, Maraffi T, Mercat A, Rodriguez PO, Shahin J, Sibley S, Spadaro S, Vaporidi K, Wilcox ME, Brochard L; Canadian Critical Care Trials Group and; REVA Network. Study protocol for a randomized controlled trial of Proportional Assist Ventilation for Minimizing the Duration of Mechanical Ventilation: the PROMIZING study. Trials. 2023 Mar 27;24(1):232. doi: 10.1186/s13063-023-07163-w. PMID 36973743
- See also: Published Protocol — https://promizingstudy.com/wp-content/uploads/2023/03/Trials-Promizing.pdf
- See also: The PROMIZING trial enrollment algorithm for early identification of patients ready for unassisted breathing — https://ccforum.biomedcentral.com/articles/10.1186/s13054-022-04063-4
- See also: PROMIZING Website — https://promizingstudy.com/

DOCUMENTS (3):
  • Study Protocol (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT02447692/Prot_003.pdf
  • Statistical Analysis Plan: Original (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT02447692/SAP_005.pdf
  • Statistical Analysis Plan: Updated (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT02447692/SAP_006.pdf